CLINICAL TRIAL: NCT06391502
Title: Effect of Multi-component Exercise Intervention Program on the Degree of Frailty in Hospitalized Patients After Venous Hemolysis in Acute Ischemic Stroke
Brief Title: Vivifrail Program on the Degree of Debilitation in Hospitalized Patients After Venous Hemolysis in Acute Ischemic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: zhangxuemei
Record Dates: First submitted 2024-01-07; First posted 2024-04-30 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-04

CONDITIONS: Ischemic Stroke; Exercise Therapy; Frailty
MeSH Terms: conditions — Ischemic Stroke; Frailty

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine exercise group (No Intervention): The routine exercise care group, that is, the control group, will complete the routine exercise care of patients with acute ischemic stroke after venous hemolytic surgery in accordance with the hospital regulations: From 24 hours after surgery, patients with mild and moderate stroke can be turned over in bed (once every 2 hours), ankle pump exercise (three times a day), and transitional bedside rehabilitation exercise (such as walking around the bed, etc.) after no discomfort.
- Multicomponent exercise group (Experimental): Select the corresponding intervention according to the SPPB score:0-3 scores (Plan A) :1. Walking 2.Relax your hand 3.Lift a bottle 4.Leg extensions with an ankle weight 5.Getting up from a chair with help 6.Holding onto the person who helps you 7.Arm stretching 4-6 scores(Plan B):1. Walking 2.Lift a bottle 3.Squeeze a ball 4.pretend to sit 5.Walking on tip toes and heels 6.Arm stretching in a chair 7.Stretch your arms up with your hands clasped;7-9 scores(Plan C):1.Walking 2.Roll-up a small towel 3.Take two plastic bottles filled with 500ml of water 4.Getting up from a chair 5.Walking over obstacles 6.Walking in a figure of eight 7.Leg stretching sit in a chair 8.Arm stretching;10-12 scores( Plan D):1.Walking 2.Twist a towel 3.Lift a bottle 4.Getting up from a chair 5.Going up and down stairs 6.Walking in a figure of eight 7.Walking while touching a balloon 8.Arm stretching;See details at http://vivifrail.com/
  Interventions: Behavioral: Multi-component Exercise Intervention Program

INTERVENTIONS:
Behavioral: Multi-component Exercise Intervention Program — The Vivifrail program (http://vivifrail.com) is a home-based exercise program that focuses on personalized multi-component exercise prescriptions based on an elderly person's functional abilities, including resistance/strength, balance, flexibility, and cardiovascular endurance exercise (i.e., walking).
  During hospitalization, patients who meet the criteria of sodium intake will be screened, and then divided into groups according to the method of randomized controlled trial. The experimental group will carry out corresponding exercise plan according to the results of SPPB.
  Arms: Multicomponent exercise group

SUMMARY:
Physical exercise is an effective strategy to maintain functional ability and improve debilitating symptoms in the elderly.In addition to functional enhancement, exercise is considered a cornerstone for enhancing cognitive function in debilitated older adults with cognitive impairment and dementia.The investigators evaluated the effect of the Vivifrail exercise intervention on the degree of debilitation in elderly hospitalized patients after venous hemolysis in acute ischemic stroke

DETAILED DESCRIPTION:
Elderly patients who are acutely hospitalized, including those who are able to walk independently, spend most of their stay in bed.In addition to worsening their functional status leading to significant muscle wasting and the development of other symptoms, it also increases the risk of cognitive decline and dementia in older adults, which is more pronounced in patients with acute ischemic stroke after venous hemolysis, and increases awareness of the need to replace prolonged bed rest with physical activity or exercise.Because there is evidence that this therapy during hospitalization is effective;A large number of studies have shown that rehabilitation training for AIS patients within 24 hours of onset is beneficial food.

In addition, exercise can reduce the damage caused by acute illness and hospitalization.Even so, it has not been established whether exercise therapy affects the degree of weakness or whether weakness affects response to treatment.

While frailty is not a disease, it can affect the presentation of many age-related diseases and the response to treatment.For example, after a short period of strength exercise in frail elderly people, autophagy in muscle cells is activated, affecting the overall health of the muscles and thus the ability to move.Similarly, the inflammatory response increases after vigorous aerobic exercise.It was also less clear whether individuals with higher frailty had any response to the intervention.

Multi-Component Exercise（Vivifrail） is an innovative multi-component exercise program that includes strength training, endurance training, balance training, and flexibility training to improve the exerciser's gait, balance, and cardiorespiratory function by increasing muscle mass, strength, and endurance.Recent studies have shown that it is one of the best ways to improve patients' gait, balance, cardiopulmonary function and cognitive executive function, as well as the best way to treat frailty, and can reduce the risk of falls and delay cognitive decline in elderly hospitalized patients with neurocognitive disorders.

The objective of this study was to examine the effect of exercise intervention on the level of frailty in older adults admitted for venous hemolysis for acute ischemic stroke.The effects of baseline frailty levels on the intervention, effectiveness of frailty, changes in Physical function (Modified Barthel Index (MBI), Short Physical Performance Battery (SPPB), and other health outcomes were determined.

ELIGIBILITY:
Inclusion Criteria:

1. Over 65 years of age;
2. Hospitalized patients diagnosed with ischemic stroke;
3. barthel index ≥60;
4. Muscle strength of both upper and lower limbs is above grade 3;
5. The pre-frailty and frailty state of the modified 5 Frailty Index (mFI-5) standard;
6. Patients willing to cooperate and sign informed consent

Exclusion Criteria:

1. fracture (within three months),
2. severe cognitive impairment, or severe dementia;
3. unable or unwilling to cooperate, any other unstable medical condition, or conditions that would prevent physical activity

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery（SPPB） | This outcome measure will be assessed within the first 2 days（Day 2） and at 1 month（Month 1） after intravenous thrombolysis in acute ischemic stroke.
  The SPPB test to determine the level of frailty is a composite of the following three separate measures:
  1. - Balance test.
  2. - Walking speed test over 4 meters.
  3. - Test of getting up from a chair. Add the points of the SPPB test (1 to 3) to determine the grade.
     * If due to limitations, you have not performed the SPPB test and you have elected to use the 6-meter walking test, the following values will be used to recommend the physical exercise program. Points 0-3 scores are considered as disability and given program A intervention; A score of 4-6 is considered as the early stage of asthenia and B intervention program is given; A score of 7-9 was considered as weak and C intervention program was given; A score of 10-12 is considered as healthy people and D intervention program is given
Modified Barthel Index | This outcome measure will be assessed within the first 2 days（Day 2） and at 1 month（Month 1） after intravenous thrombolysis in acute ischemic stroke.
  The assessment of the individual's daily living ability includes 10 items, including eating, decoration, bathing, etc. Each index is divided into 5 levels: complete dependence, greater dependence, medium dependence, lesser dependence, and independence. The higher the score, the better the independence of daily life, a total of 100 points
FRAIL Scale | This outcome measure will be assessed within the first 2 days（Day 2） and at 1 month（Month 1） after intravenous thrombolysis in acute ischemic stroke.
  Including fatigue, can not go up a flight of stairs, can not walk 500 m, suffering from more than 5 diseases, body mass decline a total of 5 indicators, using two classification scoring method, a total of 5 points.
  0 was classified as no frailty, 1-2 as pre-frailty, and ≥3 as frailty.
Grip | This outcome measure will be assessed within the first 2 days（Day 2） and at 1 month（Month 1） after intravenous thrombolysis in acute ischemic stroke.
  Use electronic grip dynamometer (Model:
  EH101) Before measurement, the instrument was calibrated to 0, the grip distance was adjusted, the fingers were naturally placed in the grip groove position, the study subjects were seated in the end position, the arm extension did not exceed 30 degrees, the upper arm and the forearm were 90 degrees, and the hands were measured with the maximum strength, the measurement interval was about 1 minute, so that the measuring hand could have enough relaxation and rest. A total of three tests were conducted.
  Average the ultimate grip strength, accurate to 0.1kg.

SECONDARY OUTCOMES:
Patient Health Questionaire - 9 items，PHQ -9 | This outcome measure will be assessed within the first 2 days（Day 2） and at 1 month（Month 1） after intravenous thrombolysis in acute ischemic stroke.
  It included 9 symptom scales and 1 overall functional assessment. Symptom scales were evaluated as follows: loss of interest, low mood, sleep disorders, fatigue, eating disorders, inferiority, difficulty in concentration, psychomotor delay, suicide symptoms, and item 10 was the overall functional assessment.
  The item definition was expressed in the form of short sentences, with a 4-level score ranging from 0 to 3, and the frequency of symptom occurrence in nearly 2 weeks.
  (0 indicates no symptoms, 1 indicates several days of symptoms, 2 indicates more than 7 days of symptoms, and 3 indicates almost every day of symptoms), the overall functional evaluation item is rated according to the degree of impact of symptoms on work, family or social function (0 indicates no, 1 indicates some impact, 2 indicates very impact, and 3 indicates very impact).
HendrichⅡfall risk model,HFRM | Acute ischemic stroke was evaluated within 48h of intravenous thrombolysis up to 4 weeks.
  There were 8 items including male, depressive state, dizziness, taking anti-epileptic drugs, standing up and walking test, and confusion. The total score was 16 points, and ≥5 was classified as high risk

CONTACTS AND LOCATIONS:
Overall Officials: xuemei zhang, master, Study Chair — Affiliated Hospital of Nantong University
Locations (1):
- AHNantongU, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Exercise Intervention protocols

REFERENCES:
- [Result] Martinez-Velilla N, Casas-Herrero A, Zambom-Ferraresi F, Saez de Asteasu ML, Lucia A, Galbete A, Garcia-Baztan A, Alonso-Renedo J, Gonzalez-Glaria B, Gonzalo-Lazaro M, Apezteguia Iraizoz I, Gutierrez-Valencia M, Rodriguez-Manas L, Izquierdo M. Effect of Exercise Intervention on Functional Decline in Very Elderly Patients During Acute Hospitalization: A Randomized Clinical Trial. JAMA Intern Med. 2019 Jan 1;179(1):28-36. doi: 10.1001/jamainternmed.2018.4869. PMID 30419096
- [Result] Casas-Herrero A, Saez de Asteasu ML, Anton-Rodrigo I, Sanchez-Sanchez JL, Montero-Odasso M, Marin-Epelde I, Ramon-Espinoza F, Zambom-Ferraresi F, Petidier-Torregrosa R, Elexpuru-Estomba J, Alvarez-Bustos A, Galbete A, Martinez-Velilla N, Izquierdo M. Effects of Vivifrail multicomponent intervention on functional capacity: a multicentre, randomized controlled trial. J Cachexia Sarcopenia Muscle. 2022 Apr;13(2):884-893. doi: 10.1002/jcsm.12925. Epub 2022 Feb 11. PMID 35150086
- [Result] Perez-Zepeda MU, Martinez-Velilla N, Kehler DS, Izquierdo M, Rockwood K, Theou O. The impact of an exercise intervention on frailty levels in hospitalised older adults: secondary analysis of a randomised controlled trial. Age Ageing. 2022 Feb 2;51(2):afac028. doi: 10.1093/ageing/afac028. PMID 35180287
- [Result] Martinez-Velilla N, Casas-Herrero A, Zambom-Ferraresi F, Suarez N, Alonso-Renedo J, Contin KC, de Asteasu ML, Echeverria NF, Lazaro MG, Izquierdo M. Functional and cognitive impairment prevention through early physical activity for geriatric hospitalized patients: study protocol for a randomized controlled trial. BMC Geriatr. 2015 Sep 15;15:112. doi: 10.1186/s12877-015-0109-x. PMID 26374430
- [Result] Casas-Herrero A, Anton-Rodrigo I, Zambom-Ferraresi F, Saez de Asteasu ML, Martinez-Velilla N, Elexpuru-Estomba J, Marin-Epelde I, Ramon-Espinoza F, Petidier-Torregrosa R, Sanchez-Sanchez JL, Ibanez B, Izquierdo M. Effect of a multicomponent exercise programme (VIVIFRAIL) on functional capacity in frail community elders with cognitive decline: study protocol for a randomized multicentre control trial. Trials. 2019 Jun 17;20(1):362. doi: 10.1186/s13063-019-3426-0. PMID 31208471
- [Result] Carli F, Bousquet-Dion G, Awasthi R, Elsherbini N, Liberman S, Boutros M, Stein B, Charlebois P, Ghitulescu G, Morin N, Jagoe T, Scheede-Bergdahl C, Minnella EM, Fiore JF Jr. Effect of Multimodal Prehabilitation vs Postoperative Rehabilitation on 30-Day Postoperative Complications for Frail Patients Undergoing Resection of Colorectal Cancer: A Randomized Clinical Trial. JAMA Surg. 2020 Mar 1;155(3):233-242. doi: 10.1001/jamasurg.2019.5474. PMID 31968063
- [Result] Izquierdo M. [Multicomponent physical exercise program: Vivifrail]. Nutr Hosp. 2019 Jul 1;36(Spec No2):50-56. doi: 10.20960/nh.02680. Spanish. PMID 31189323
- [Result] Sanchez-Sanchez JL, de Souto Barreto P, Anton-Rodrigo I, Ramon-Espinoza F, Marin-Epelde I, Sanchez-Latorre M, Moral-Cuesta D, Casas-Herrero A. Effects of a 12-week Vivifrail exercise program on intrinsic capacity among frail cognitively impaired community-dwelling older adults: secondary analysis of a multicentre randomised clinical trial. Age Ageing. 2022 Dec 5;51(12):afac303. doi: 10.1093/ageing/afac303. PMID 36580558
- [Result] Courel-Ibanez J, Pallares JG, Garcia-Conesa S, Buendia-Romero A, Martinez-Cava A, Izquierdo M. Supervised Exercise (Vivifrail) Protects Institutionalized Older Adults Against Severe Functional Decline After 14 Weeks of COVID Confinement. J Am Med Dir Assoc. 2021 Jan;22(1):217-219.e2. doi: 10.1016/j.jamda.2020.11.007. Epub 2020 Dec 6. No abstract available. PMID 33296679
- [Result] Izquierdo M, Rodriguez-Manas L, Sinclair AJ. Editorial: What Is New in Exercise Regimes for Frail Older People - How Does the Erasmus Vivifrail Project Take Us Forward? J Nutr Health Aging. 2016;20(7):736-7. doi: 10.1007/s12603-016-0702-5. No abstract available. PMID 27499307
- [Result] Sanchez-Sanchez JL, Udina C, Medina-Rincon A, Esbri-Victor M, Bartolome-Martin I, Moral-Cuesta D, Marin-Epelde I, Ramon-Espinoza F, Latorre MS, Idoate F, Goni-Sarries A, Martinez-Martinez B, Bonet RE, Librero J, Casas-Herrero A. Effect of a multicomponent exercise program and cognitive stimulation (VIVIFRAIL-COGN) on falls in frail community older persons with high risk of falls: study protocol for a randomized multicenter control trial. BMC Geriatr. 2022 Jul 23;22(1):612. doi: 10.1186/s12877-022-03214-0. PMID 35870875